CLINICAL TRIAL: NCT02801916
Title: Effect of Consuming Oat Bran Mixed in Water Before a Meal on Glycemic Responses in Healthy Humans - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GIL1527b
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Glucose Intolerance
Keywords: Humans; Glycemic response; Oat beta-glucan
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study subjects (Other): Each healthy subject will receive each of the interventions in randomized order.
  Interventions: Other: 0 grams oat bran; Other: 4.5 grams oat bran; Other: 13.6 grams oat bran; Other: 27.3 grams oat bran

INTERVENTIONS:
Other: 0 grams oat bran — 200 milliliters water plus 0 grams OatWell22, a commercial oat bran product containing 22% oat beta-glucan, followed by 119 grams white bread
Other: 4.5 grams oat bran — 200 milliliters water plus 4.5 grams OatWell22, a commercial oat bran product containing 22% oat beta-glucan, followed by 119 grams white bread
Other: 13.6 grams oat bran — 200 milliliters water plus 13.6 grams OatWell22, a commercial oat bran product containing 22% oat beta-glucan, followed by 119 grams white bread
Other: 27.3 grams oat bran — 200 milliliters water plus 27.3 grams OatWell22, a commercial oat bran product containing 22% oat beta-glucan, followed by 119 grams white bread

SUMMARY:
Viscous dietary fibers including oat β-glucan are one of the most effective classes of functional food ingredients for reducing postprandial blood glucose. The mechanism of action is thought to be via an increase in viscosity of the stomach contents that delays gastric emptying and reduces mixing of food with digestive enzymes, which, in turn, retards glucose absorption. Previous studies suggest that taking viscous fibers separate from a meal may not be effective in reducing postprandial glycemia. The purpose of this study is to re-assess the effect of consuming a preload of a commercially available oat-bran (4.5, 13.6 or 27.3 g) containing 22% of high molecular weight oat β-glucan (O22) mixed in water before a test-meal of white bread on glycemic responses in 10 healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Pregnancy
* Diabetes
* Recent medical or surgical hospitalization
* Use of drugs influencing glucose metabolism
* Use of drugs influencing gastrointestinal function
* Allergy to oats or wheat

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Glucose AUC | 0 to 2 hours after test meal
  Incremental area under the blood glucose response curve from 0 hours (fasting) to 2 hours after eating ignoring area below fasting

SECONDARY OUTCOMES:
Peak rise of blood glucose | 0 to 2 hours after test meal
  Highest concentration of blood glucose within 2 hours of eating minus the fasting glucose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc

IPD SHARING:
Plan to Share IPD: No